CLINICAL TRIAL: NCT06810869
Title: Exploratory Clinical Study on Induced Pluripotent Stem Cell Derived Exosomes (iPSC-Exos) for the Treatment of Stable Vitiligo
Brief Title: Induced Pluripotent Stem Cell Derived Exosomes Nasal Drops for the Treatment of Stable Vitiligo
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Wannan Medical College (Other)
Collaborators: Guidon Pharmaceutics Ltd. (Industry)
Responsible Party: Principal Investigator, Ruzhi Zhang, MD; PhD, Second Affiliated Hospital of Wannan Medical College
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WYEFYLS2024121
Record Dates: First submitted 2025-01-22; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Stable Vitiligo
Keywords: iPSC; exosome; Stable Vitiligo
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exosomes group (Experimental): group1-low-dose group, 3 patients will receive doses of GD-iExo-003 at 1×10^8 particles per 4 square centimeters of lesion area in 100 μL. group2-mid-dose group, 3 patients will receive doses of GD-iExo-003 at 3×10^8 particles per 4 square centimeters of lesion area in 100 μL. group3-high-dose group, 3 patients will receive doses of GD-iExo-003 at 9×10^8 particles per 4 square centimeters of lesion area in 100 μL. The administration method is microneedle injection, with each injection being 100 ul. Once every 2 weeks, for a total treatment duration of 3 months, with an additional follow-up period of 6 months
  Interventions: Drug: human induced pluripotent stem cell derived exosomes （GD-iExo-003）
- placebo group (Placebo Comparator): Patients in this arm will be given a placebo. The administration method is microneedle injection, with each injection being 100 ul. Once every 2 weeks, for a total treatment duration of 3 months, with an additional follow-up period of 6 months.
  Interventions: Drug: a placebo of exosomes derived from human induced pluripotent stem cell for injection

INTERVENTIONS:
Drug: human induced pluripotent stem cell derived exosomes （GD-iExo-003） — human induced pluripotent stem cell derived exosomes （GD-iExo-003）
  Arms: Exosomes group
Drug: a placebo of exosomes derived from human induced pluripotent stem cell for injection — a placebo of exosomes derived from human induced pluripotent stem cell for injection
  Arms: placebo group

SUMMARY:
Evaluate the efficacy of induced pluripotent stem cell-derived exosomes (iPSC-Exos) for the treatment of stable vitiligo

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy and safety of iPSC-Exos in the treatment of localized stable vitiligo. iPSC-Exos have been found to possess the ability to promote cell survival, proliferation, and repair, potentially improving skin pigmentation in vitiligo patients by modulating the survival and function of melanocytes.

This study will consist of 2 parts, with part 1 being a dose-escalation study and part 2 being an expanded safety study based on part 1 findings.

A traditional 3+3 dose escalation design will be implemented in part 1. Cohort 1: receive 1×10^8 particles per time; cohort 2: 3×10^8 particles per time and cohort 3: 9×10^8 particles per time.

In part 2, 20 subjects will be randomized in a 1:1 ratio [exosome (n=10) or exosome placebo (n=10)]. The dose level will be determined by Data Safety Monitoring Board based on part 1.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the trial treatment protocol and visit schedule, voluntarily enroll in the study, and provide written informed consent;
2. Aged 18-60 years old (inclusive of 18 and 60 years);
3. Clinically diagnosed with stable localized vitiligo (in accordance with the 2021 Consensus on the Diagnosis and Treatment of Vitiligo); Stability criteria: ① A score of 0 on the Vitiligo Disease Activity (VIDA) scale; ② Clinical characteristics: white patches appear porcelain white, with clear or pigmented edges; ③ No Koebner phenomenon (for ≥1 year); ④ Wood's lamp examination: lesions appear white with clear boundaries, and the area under Wood's light is ≤ visual estimation area, indicating stability. Skin CT and dermatoscopy images may also be referenced for diagnostic assistance. Localization criteria: Refers to single lesions, with an area classified as grade 1 (lesion area <1% of total body surface area), where it is not yet possible to determine whether the presentation is segmental or non-segmental at the time of consultation.
4. Lesions have been stable for more than 6 months, with a number of foci ≥3, ensuring that at least 2 lesions have an area >2cm²;
5. Have no plans for conception during the study period and for 3 months after the last administration, and can adopt effective contraceptive measures;
6. Agree to suspend any other anti-vitiligo treatments outside of the study protocol during participation in this clinical research (excluding cosmetic cover-ups).

Exclusion Criteria:

1. Individuals with clinically significant multiple or severe drug allergies, or those who have had serious allergic reactions to treatments, or where the investigator anticipates that the participant may be allergic to the study medication or any of its components;
2. Participants diagnosed with progressive vitiligo or moderate-to-severe stable vitiligo;
3. Total depigmented area ≥1% of body surface area (BSA);
4. Those who have received other treatments for vitiligo within the recent past (within 3 months), such as corticosteroids, JAK inhibitors, topical herbal medicines, depigmentation therapy, melanocyte-keratinocyte transplant surgery, phototherapy, etc.;
5. Participants with other active pigmented skin diseases during the screening period, such as pityriasis alba, senile leukoderma, chemical/drug-induced vitiligo, hyperpigmentation due to malignancy, post-inflammatory hyperpigmentation, ataxia telangiectasia, tuberous sclerosis, melasma, congenital hypopigmentation disorders, etc.;
6. Evidence of active inflammatory skin disease or skin condition during the screening period, such as atopic dermatitis, psoriasis, discoid lupus, leprosy, syphilis, seborrheic dermatitis, etc., which the investigator assesses might interfere with the evaluation of response and safety regarding vitiligo treatment;
7. Pregnant or breastfeeding women;
8. Participants with a history or current diagnosis of other autoimmune diseases and major illnesses: tuberculosis, AIDS, malignancies, cardiovascular and cerebrovascular diseases, liver and kidney diseases, etc.;
9. Individuals with a history of substance or alcohol abuse or those suffering from mental health conditions;
10. Abnormal blood test results that the investigator judges could affect the assessment of efficacy and safety of the participant or the trial outcomes;
11. Any other circumstances where the investigator believes that the participant's compliance may be affected or they are unsuitable to participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-02-05 (Estimated); Primary Completion 2026-11-17 (Estimated); Study Completion 2026-11-17 (Estimated)

PRIMARY OUTCOMES:
adverse events as assessed by CTCAE | Screening and 1 day, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks, 14 weeks，18 weeks，22 weeks，24 weeks after the first injection
  all potentially treated subjects to assess the safety

SECONDARY OUTCOMES:
Local Adverse Reactions | Screening and 1 day, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks, 14 weeks，18 weeks，22 weeks，24 weeks after the first injection
  Changes in the lesions at the site of the white patches after treatment, such as erythema, blisters, erosion, scaling, pigmentation, Koebner phenomenon, etc
Systemic Adverse Reactions | Screening and 1 day, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks, 14 weeks，18 weeks，22 weeks，24 weeks after the first injection
  blood tests to check liver function indicators-Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST)-and kidney function indicators-Creatinine (Cr), Blood Urea Nitrogen (BUN)
Changes in the area of white patches | Screening and 1 day, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks, 14 weeks，18 weeks，22 weeks，24 weeks after the first injection
  Using the grid counting method to calculate the area of white patches
Vitiligo Area Scoring Index (VASI) change | Screening and 1 day, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks, 14 weeks，18 weeks，22 weeks，24 weeks after the first injection
  VASI = Number of Hand Palm Units × Percentage of Depigmentation, with VASI values ranging from 0 to 100. One palm area is divided into 32 finger-joint units, where the palm center area accounts for 18 finger-joint units representing 0.54%, and one finger-joint unit represents 0.03%.
  VASI Improvement Rate = (VASI score before treatment - VASI score after treatment) / VASI score before treatment × 100%. VASI50 is defined as an improvement in the VASI score of ≥50% from baseline; VASI75 is defined as an improvement in the VASI score of ≥75% from baseline.
Vitiligo Noticeability Scale (VNS) change | Screening and 1 day, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks, 14 weeks，18 weeks，22 weeks，24 weeks after the first injection
  This questionnaire includes assessments of appearance noticeability and psychosocial impact, with higher scores indicating a greater level of impact.
Dermatology Life Quality Index (DLQI) change | Screening and 1 day, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks, 14 weeks，18 weeks，22 weeks，24 weeks after the first injection
  The questionnaire contains 10 questions, with each option scored from 0 to 3. If a question is not relevant, it is also scored as 0. The score range is from 0 to 30, with higher scores indicating a greater impact on the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Wannan Medical College, Wuhu, Anhui, China

IPD SHARING:
Plan to Share IPD: No
The study will not share individual participant data to other researchers.